CLINICAL TRIAL: NCT00002826
Title: A PILOT PHASE II TRIAL OF PSC 833 MODULATION OF MULTIDRUG RESISTANCE TO PACLITAXEL IN THE TREATMENT OF METASTATIC CARCINOMA OF THE BREAST
Brief Title: Drug Resistance Inhibition in Treating Women With Recurrent or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065011; E-1195
Record Dates: First submitted 1999-11-01; First posted 2004-05-12 (Estimated); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; valspodar

INTERVENTIONS:
Drug: paclitaxel
Drug: valspodar

SUMMARY:
RATIONALE: Some tumors become resistant to chemotherapy drugs. Combining PSC 833 with a chemotherapy drug may reduce resistance to the drug, and allow the tumor cells to be killed.

PURPOSE: Phase II trial to study the effectiveness of PSC 883 and paclitaxel in treating women who have recurrent or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the antitumor activity, as measured by frequency of objective response and time to progression, of the multidrug resistance modulator PSC 833 in combination with paclitaxel in women with recurrent or metastatic breast cancer. II. Describe the toxicity of this regimen.

OUTLINE: All patients receive PSC 833 by mouth every 6 hours for a total of 12 doses. Paclitaxel is infused over 3 hours, after the 5th dose of PSC 833. Treatment is repeated every 3 weeks in stable and responding patients. PSC 833 must not be mixed with grapefruit juice. Growth factors may be used at the discretion of the investigator. Patients are followed every 3 months for the first two years, then every 6 months for years 2-5, and then annually thereafter.

PROJECTED ACCRUAL: It is anticipated that approximately 36 patients will be entered over 24 months if there are at least 6 responses in the first 17 patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed adenocarcinoma of the breast that is recurrent or metastatic No CNS metastases Bidimensionally measurable disease required Patients with bone sites only are not eligible Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 and over Sex: Women only Menopausal status: Not specified Performance status: ECOG 0-2 Hematopoietic: Platelet count at least 100,000/mm3 Absolute granulocyte count at least 1,500/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL AST less than 2.5 times upper limit of normal Renal: Creatinine no greater than twice upper limit of normal Other: No allergy to cyclosporine or to drugs formulated with Cremophor (e.g., some anesthetics and muscle relaxants) No active unresolved infection More than 7 days since parenteral antibiotics No second malignancy within 5 years except: In situ cervical cancer Nonmelanomatous skin cancer No pregnant or nursing women Adequate contraception required of fertile women

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Prior anthracyclines or medical contraindication to anthracycline therapy required No prior paclitaxel or taxotere No more than 1 prior regimen for metastatic or recurrent disease Adjuvant chemotherapy within 6 months of diagnosis of metastatic disease considered therapy for advanced disease At least 3 weeks since chemotherapy Endocrine therapy: At least 3 weeks since hormonal therapy for metastases Radiotherapy: Not specified Surgery: Not specified Other: No concurrent treatment with any of the following agents proven to affect blood levels of cyclosporine: Diltiazem Nicardipine Verapamil Fluconazole Itraconazole Ketoconazole Clarithromycin Erythromycin Methylprednisolone Prednisolone Allopurinol Bromocriptine Danazol Metoclopramide Nafcillin Rifampin Carbamazepine Phenobarbital Phenytoin Octreotide Ticlopidine

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 1997-08-14 (Actual); Primary Completion 2003-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert W. Carlson, MD, Study Chair — Stanford University
Locations (9):
- United States (9):
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - Stanford University Medical Center, Stanford, California
  - Hunterdon Regional Cancer Program, Flemington, New Jersey
  - Kimball Medical Center, Lakewood, New Jersey
  - Fox Chase Cancer Center at Virtua-Memorial Hospital Burlington County, Mount Holly, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - St. Francis Medical Center, Trenton, New Jersey
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Carlson RW, O'Neill A, Goldstein L, et al.: A phase II trial of PSC-833 modulation of multidrug resistance to paclitaxel in breast cancer: a pilot trial of the Eastern Cooperative Oncology Group. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-234, 2002.